CLINICAL TRIAL: NCT03160612
Title: Investigation of the Effects of Independent Transfer Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Boninger, Professor and UPMC Endowed Vice Chair for Research, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15030691; H133N110011 (Other Grant/Funding Number: U.S. Department of Education)
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Wheelchair Transfers
Keywords: Wheelchair; Biomechanics; Transfer; Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Other): Transfer Training Subjects will be randomized to receive the transfer training either after baseline measures are collected (case) during visit 1.
  Interventions: Behavioral: Transfer Training
- Control (Other): Transfer Training Subjects will be randomized to receive the transfer training during the follow-up testing at visit 2.
  Interventions: Behavioral: Transfer Training

INTERVENTIONS:
Behavioral: Transfer Training — Transfer training interventions will take approximately 1 hour to complete and consist of an interactive web based module that participants interact with which includes text, pictures, videos and time to practice new skills. Additionally, participants will receive an educational handout summarizing the online module.

SUMMARY:
The objective of this research study is to 1) evaluate the effectiveness of web based transfer training materials for wheelchair users and 2) determine the reliability of a refined transfer assessment instrument (TAI) as completed by individuals who use wheelchairs for a majority of mobility and clinicians who score transfers in-person and remotely.

DETAILED DESCRIPTION:
Up to 125 participants will be recruited for this study. Investigators will recruit individuals who use a wheelchair for a majority of mobility (>40 hours per week), who are over 18 years old, who do not have a history of heart or lung conditions that could become worse with up to 6 back and forth transfers to a mat table, and who can independently transfer to and from a surface within 30 seconds without use of their legs.

This study will require two visits that will take approximately 2 hours total to complete. Subjects will be asked to fill out a series of questionnaires so that investigators can collect demographic information (i.e. age, race, diagnosis, date of diagnosis, handedness, and preferred leading arm for transfers), their weight, and information about arm pain. Physical exams qualifying shoulder and wrist pathology will also be completed. Subjects will then be asked to perform up to six back and forth transfers to a mat table.

Following this, subjects will be randomized into two groups; one group that will receive transfer training immediately, and one group that will receive the transfer training after the follow up visit (control).

Subjects in the immediate transfer training group will receive training about about proper transfer techniques. After training, they will then complete the repeated transfer portion of the protocol a second time. Subjects will be instructed to practice the new skills they learned and then return within 7 days to complete only the repeated transfer portion of the protocol.

Subjects in the delayed transfer training group will be instructed to return within 7 days. Subjects will complete the repeated transfer portion of the protocol a second time. Subjects will then receive training about proper transfer techniques and after complete the repeated transfer portion of the protocol a third time.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Utilizes a wheelchair for the majority of mobility (over 40 hours per week)
3. Ability to transfer independently (may use equipment)
4. Self-report ability to complete a transfer to and from a surface in 30 seconds
5. English speaking

Exclusion Criteria:

1. Current or recent history (last 3 months) of pressure sores that may be exacerbated by multiple transfers
2. Active use of the lower limb muscles during transfers
3. Upper extremity pain that inhibits the ability to perform transfers or bear weight on the upper extremities
4. Other neurologic condition that could impair learning
5. History of heart or lung conditions that would be made worse by completing up to six back and forth transfers to a mat table

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07-02 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Change in Transfer Assessment Instrument (TAI) Scores | Baseline visit and visit 2 (which will occur within 7 days of baseline)
  Transfer assessment instrument (TAI) scores will be collected both before and after the training to assess for changes in the score.

SECONDARY OUTCOMES:
Shoulder pain | Baseline visit
  A physical exam will be performed to qualify shoulder pain.
Shoulder pathology | Baseline Visit
  A physical exam will be performed to qualify shoulder pathology.
Wrist Pain | Baseline visit
  A physical exam will be performed to qualify wrist pain.
Wrist pathology | Baseline Visit
  A physical exam will be performed to qualify wrist pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boninger, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.